CLINICAL TRIAL: NCT02118597
Title: Non-interventional Study to Observe Triple Combination Therapy With Boceprevir or Simeprevir Plus Peginterferon Alfa-2a Plus Ribavirin for Re-treatment of Chronic Hepatitis C in Hungary (IMPERIAL)
Brief Title: An Observational Study Examining the Use of Triple Combination Therapy With Boceprevir, Peginterferon Alfa-2a and Ribavirin in the Re-Treatment of Chronic Hepatitis C Patients
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to the Sponsor's decision.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29278
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum used to analyze levels of hepatitic c virus (HCV) ribonucleic acid (RNA)

GROUPS / COHORTS (1):
- Triple Combination Therapy: Participants who demonstrated genotype 1 chronic hepatitis C infection and had a history of unsuccessful treatment with pegylated interferon (peginterferon) alfa + ribavirin, and who were subjected to receive a triple combination therapy with simeprevir or boceprevir plus peginterferon alfa-2a and ribavirin were observed.
  Interventions: Drug: Boceprevir; Drug: Simeprevir; Drug: Pegylated Interferon (Peginterferon) Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir — Boceprevir administered according to corresponding summary of product characteristics (SmPC).
  Other Names: Victrelis
Drug: Simeprevir — Simeprevir administered according to corresponding summary of product characteristics (SmPC).
  Other Names: Olysio
Drug: Pegylated Interferon (Peginterferon) Alfa-2a — Pegylated interferon (peginterferon) alfa-2a according to corresponding summary of product characteristics (SmPC).
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin according to corresponding summary of product characteristics (SmPC).
  Other Names: Copegus

SUMMARY:
This prospective, national, multicenter, non-interventional study examined the use of triple combination therapy with boceprevir, pegylated interferon (peginterferon) alfa-2a and ribavirin in re-treating participants with genotype 1 chronic hepatitis C (CHC) infection. Dosing and treatment duration were at the discretion of the investigator in accordance with local clinical practice and local labeling. Participants were to be observed for the duration of their triple combination therapy and for up to 24 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Genotype 1 CHC infection
* Prior unsuccessful treatment with peginterferon alfa plus ribavirin (null-response, partial response and relapsed participants)
* Receiving triple combination therapy with boceprevir, peginterferon alfa-2a and ribavirin according to standard of care and in line with local labeling
* Enrollment in the study no later than 4 weeks after start of triple combination therapy (including peginterferon alfa-2a and ribavirin lead-in phase)

Exclusion Criteria:

* Naïve participants not responding to peginterferon alfa plus ribavirin at week 4 (HCV RNA drop < 1 log10) or at week 12 (HCV RNA >/= 15 international units/milliliter [IU/mL]) and switching to triple combination therapy with boceprevir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with genotype 1 chronic hepatitis C (CHC) infection taking triple combination therapy (boceprevir, peginterferon alfa-2a and ribavirin)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Hungary (6):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Eger
  - Kaposvár
  - Szombathely

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 participants were enrolled in 8 study centers.
Groups:
- Triple Combination Therapy: Participants with genotype 1 chronic hepatitis C infection and a history of unsuccessful treatment with pegylated interferon (peginterferon) alfa plus ribavirin, who received a triple combination therapy with boceprevir plus peg-interferon alfa-2a plus ribavirin, were observed.
Period: Overall Study
Arm/Group | Triple Combination Therapy
Started | 19
Completed | 3
Not Completed | 16
Not completed — Sponsor terminated the study | 14
Not completed — Serious Adverse Event | 1
Not completed — Investigator's decision | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.73 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response 24 (SVR24) Rate
Description: The SVR 24 rate is defined as percentage of participants with Hepatitis C virus (HCV) Ribonucleic Acid (RNA) less than 15 international unit/milliliter (IU/mL) after the 24-weeks follow-up.
Time Frame: 24 weeks after end of treatment (EOT) at Week 72
Population: Due to the early termination of the study follow-up of the vast majority of the participants was not possible and data were not collected. Therefore, results for this outcome measure are based on one participant.
Measure: Number; unit: percentage of participants
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 1
percentage of participants | 0

2. Secondary Outcome: Percentage of Participants With Virological Response
Description: Virological response is defined as HCV RNA <15 IU/mL.
Time Frame: Weeks 4, 8, 12, and 24
Population: Intent to treat (ITT) population included all enrolled participants. Here, 'n' indicated number of participants with virological response data at evaluated time points.
Measure: Number; unit: percentage of participants
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 19
percentage of participants
  Week 4 (n=3) | 0.0
  Week 8 (n=18) | 73.7
  Week 12 (n=17) | 73.7
  Week 24 (n=16) | 78.9

3. Secondary Outcome: Number of Participants With Virological Breakthrough
Description: Virological breakthrough is defined as either HCV RNA >=15 IU/mL in participants with prior virological response or as an increase in HCV RNA >/=1 log10 above nadir.
Time Frame: Up to Week 48
Population: ITT population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 19
participants | 1

4. Secondary Outcome: Number of Participants With Virological Relapse
Description: Virological response is defined as HCV RNA >/=15 IU/mL during the treatment free follow-up period in participants with virological response at the end of treatment.
Time Frame: Week 49 up to Week 72
Population: ITT population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 19
participants | 1

5. Secondary Outcome: Number of Participants With Treatment Discontinuation Due to Futility
Description: Treatment discontinuation due to futility is defined as HCV RNA drop <3 log10 at Week 8, HCV RNA >/=100 IU/mL at Week 12, or HCV RNA >/=15 IU/mL at Week 24.
Time Frame: Up to Week 48
Population: ITT population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 19
participants | 2

6. Secondary Outcome: Number of Participants With Treatment Discontinuation
Description: Treatment discontinuation is reported by sub-categories of reasons for treatment discontinuation. Futility rule is defined as HCV RNA drop <3 log10 at Week 8, HCV RNA >/=100 IU/mL at Week 12, or HCV RNA >/=15 IU/mL at Week 24.
Time Frame: Up to Week 48
Population: ITT population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 19
participants
  Sponsor's decision | 7
  Adverse event | 4
  Futility rule | 2

7. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 72 weeks
Population: ITT population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 19
participants | 17

8. Secondary Outcome: Percentage of Participants With Positive Predictive Value of Participant Demographics for SVR Rate
Description: Demographic characteristics recorded were age and gender. Predictive value of these characteristics for SVR rate was to be assessed.
Time Frame: Screening (before Week 1)
Population: Predictive values of participant demographics could not be analyzed as the SVR24 rate was based on one participant.
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants With Positive Predictive Value of Liver Fibrosis
Description: The following sub-categories of liver fibrosis were determined in this study: 1) no cirrhosis, 2) bridging fibrosis and 3) cirrhosis. Predictive value of these sub-categories of liver fibrosis for SVR rate was to be assessed.
Time Frame: Screening (before Week 1)
Population: Predictive values of sub-categories of liver fibrosis could not be analyzed as the SVR24 rate was based on one participant.
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 0

10. Secondary Outcome: Predictive Value of HCV Disease Characteristics
Description: HCV disease characteristics evaluated were HCV genotype (subtype), including HCV 1(a) and HCV 1(b). Predictive value of these disease characteristics for SVR rate were to be assessed.
Time Frame: Screening (before Week 1)
Population: Predictive values of HCV disease characteristics could not be analyzed as the SVR24 rate was based on one participant.
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants With Positive Predictive Value of Previous Virological Response (Null-response, Partial Response, or Relapse)
Description: Previous virological response was sub-categorized into the following categories: null-response, partial response, or relapse. Predictive value of these sub-categories for SVR rate were to be assessed.
Time Frame: Up to 72 weeks
Population: Predictive values of previous virological response could not be analyzed as the SVR24 rate was based on one participant.
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent form up to the end of study (up to 72 weeks)
Groups:
- Triple Combination Therapy: Participants who demonstrated genotype 1 chronic hepatitis C infection and had a history of unsuccessful treatment with pegylated interferon (Peg-interferon) alfa + ribavirin, and who were subjected to receive a triple combination therapy with simeprevir or boceprevir plus peg-interferon alfa-2a and ribavirin were observed.
Arm/Group | Triple Combination Therapy
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Combination Therapy (N=19)
Administration site cellulitis (Infections and infestations) | 1
Ileus (Gastrointestinal disorders) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Combination Therapy (N=19)
Influenza like illness (General disorders) | 1
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.